CLINICAL TRIAL: NCT03174197
Title: Phase I/II Study to Evaluate the Safety and Clinical Efficacy of Atezolizumab (aPDL1) in Combination With Temozolomide and Radiation in Patients With Newly Diagnosed Glioblastoma (GBM)
Brief Title: Atezolizumab in Combination With Temozolomide and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0867; NCI-2018-02629 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0867 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — atezolizumab; Radiotherapy; Radiation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adjuvant phase (temozolomide, atezolizumab) (Experimental): Patients receive temozolomide PO on days 1-5 and atezolizumab IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Temozolomide
- Concurrent phase (temozolomide, atezolizumab, RT) (Experimental): Patients receive temozolomide PO daily on days 1-42 and atezolizumab IV over 30-60 minutes on day 1, 15, 29, and 42. Patients undergo RT 5 days per week (Monday-Friday) for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Radiation: Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
  Arms: Concurrent phase (temozolomide, atezolizumab, RT)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase I/II trial studies the side effects and how well atezolizumab works in combination with temozolomide and radiation therapy in treating patients with newly diagnosed glioblastoma. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy beams to kill tumor cells and shrink tumors. It is not yet known how well atezolizumab works in combination with temozolomide and radiation therapy in treating patients with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of atezolizumab in combination with radiation and temozolomide during the concurrent stage and in combination with temozolomide during the adjuvant stage. (Phase I) II. To evaluate the overall survival (OS) of atezolizumab in combination with radiation and temozolomide and in combination with temozolomide at onset of treatment. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (ORR), duration of response, and progression free survival (PFS) of atezolizumab in combination with radiation and temozolomide during the treatment period.

CORRELATIVE OBJECTIVES:

I. Profiling tumor immune cell populations (example: immunohistochemistry [IHC] analyses of CD4, CD8, programmed death-1 [PD-1], programmed death-ligand 1 [PD-L1], and PD-L2).

II. Profiling of tumor deoxyribonucleic acid (DNA), messenger ribonucleic acid (mRNA), microRNA and epigenetic profiling (DNA methylation) and evaluation of whole exome sequencing, RNA sequencing, microRNA sequencing and cell-free circulating tumor DNA (ctDNA).

III. Peripheral blood collection for evaluation of circulating chemokines/cytokines.

OUTLINE: This is a phase I study followed by a phase II study.

PHASE I (CONCURRENT PHASE): Patients receive temozolomide orally (PO) daily on days 1-42 and atezolizumab intravenously (IV) over 30-60 minutes on day 1, 15, 29, and 42. Patients undergo radiation therapy (RT) 5 days per week (Monday-Friday) for 6 weeks in the absence of disease progression or unacceptable toxicity.

PHASE II (ADJUVANT PHASE): Patients receive temozolomide PO on days 1-5 and atezolizumab IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF).
* Ability and willingness to comply with the requirements of the study protocol.
* Have histologically confirmed World Health Organization grade IV glioma (glioblastoma or gliosarcoma). Archival tissue will be required for diagnosis confirmation. Receipt of archival tissue is not required for the start of treatment.
* Patients must have undergone surgery and must not have had any further treatment following surgery.
* Have a performance status of >= 60 on the Karnofsky performance status (KPS).
* A baseline brain magnetic resonance imaging (MRI) obtained no more than 14 days prior to study enrollment on a stable or tapering dose of steroids no greater than 4 mg a day of dexamethasone for at least 5 days.
* Patients must start treatment within 6 weeks of definitive resection.
* Absolute neutrophil count (ANC) >= 1,500 /mcL.
* Platelets >= 100,000 /mcL.
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L.
* Serum creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 x upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN.
* Serum total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN.
* International normalized ratio (INR) or prothrombin time (PT) activated partial thromboplastin time (aPTT) </=1.5 x ULN.
* All screening labs should be performed within 14 days (+ 3 working days) of treatment initiation.
* Female subject of childbearing potential should have a negative serum pregnancy test within 14 days (+ 3 working days) of study enrollment.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the duration of the study. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception during the course of the study.

Exclusion Criteria:

* Has received prior interstitial brachytherapy, implanted chemotherapy, or therapeutics delivered by local injection or convection enhanced delivery. Prior treatment with Gliadel wafers will be excluded. Prior treatment with the Optune device will be excluded.
* Is currently participating or has participated in any other newly diagnosed therapeutic trial before or after chemoradiation.
* Any serious medical condition that interferes with adherence to study procedures.
* Patients may not receive concomitant chemotherapy, hormonal therapy, immunotherapy, or radiotherapy while patients are on study.
* Malignancies other than the disease under study within 5 years prior to cycle 1, day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai Stage 0).
* Has known leptomeningeal disease, gliomatosis cerebri, extracranial disease, or multifocal disease. Subject has multifocal glioblastoma (GBM), defined as discrete sites of contrast enhancing disease without contiguous T2/fluid attenuated inversion recovery (FLAIR) abnormality that require distinct radiotherapy ports. Satellite lesions that are associated with a contiguous area of T2/FLAIR abnormality as the main lesion(s) and that are encompassed within the same radiotherapy port as the main lesion(s) are permitted.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit.
* Contraindication for undergoing MRIs.
* Inability to comply with study and follow-up procedures.
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis. Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible. Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible. Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions: Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations; rash must cover less than 10% of body surface area (BSA); disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%); no acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids).
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
* History of human immunodeficiency virus (HIV) infection or active hepatitis B (chronic or acute) or hepatitis C infection. Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible. Patients will be sampled for hepatitis B virus (HBV) deoxyribonucleic acid (DNA) and will be referred to a virologist to monitor for HBV re-activation. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA).
* Active tuberculosis.
* Severe infections within 4 weeks prior to cycle 1, day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Signs or symptoms of infection within 2 weeks prior to cycle 1, day 1.
* Received oral or IV antibiotics within 2 weeks prior to cycle 1, day 1. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Anticipation of need for a major surgical procedure during the course of the study.
* Administration of a live, attenuated vaccine within 4 weeks before cycle 1, day 1 or anticipation that such a live, attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to cycle 1, day 1 or at any time during the study and for 5 months after last dose of atezolizumab.
* Malignancies other than the disease under study within 5 years prior to cycle 1, day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g., chronic lymphocytic leukemia Rai stage 0, prostate cancer with Gleason score =< 6, and prostate-specific antigen [PSA] =< 10 mg/mL, etc.)
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway targeting agents.
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]-a or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to cycle 1, day 1.
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1. Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) (Phase I) | Up to 10 weeks
  Will monitor time to DLT continuously using a Bayesian method that assumes the median time to DLT follows an Inverse gamma distribution and that the individual times to DLT follow an exponential distribution.
Overall survival (OS) (Phase II) | Up to 3 years
  Kaplan-Meier curves will be generated for OS and median times and probabilities estimated with 95% confidence intervals.
Incidence of adverse events | Up to 3 years
  The overall toxicity rate will be estimated with exact binomial 95% confidence intervals. Adverse Events will be tabulated by grade and by their relationship to the treatment.

SECONDARY OUTCOMES:
Overall response rate | Up to 3 years
  Will be estimated with exact binomial 95% confidence intervals. Logistic regression will be used to explore the correlations between response rates and correlative markers.
Duration of response (DoR) | Up to 3 years
  Kaplan-Meier curves will be generated for DoR and median times and probabilities estimated with 95% confidence intervals.
Progression-free survival (PFS) | Up to 3 years
  Kaplan-Meier curves will be generated for PFS and median times and probabilities estimated with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Shiao-Pei S Weathers, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT03174197/ICF_000.pdf